CLINICAL TRIAL: NCT02666729
Title: Use of a Novel Contact Force Sensing Catheter for AF Ablation - Impact of TactiCath on Dormant Conduction Across the Pulmonary Veins
Acronym: FORMIDIBLE
Status: Withdrawn | Type: Observational
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: STUDY00003285
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AF Ablation Procedure: Patients with AF who are schedule for a first time pulmonary vein isolation (PVI) for AF using the TactiCath catheter. Patients will have four pulmonary veins ablated during procedure. The researcher will perform AF Ablation with contact force information on two veins. The research will perform AF Ablation without contact force information on the other two veins.
  Interventions: Procedure: AF Ablation with contact force information; Procedure: AF Ablation without contact force information

INTERVENTIONS:
Procedure: AF Ablation with contact force information — Ablation procedure will be done using TactiCath Quartz ablation catheter which can measure the amount of contact force being used. Researcher will be made aware of contact force data when performing procedure.
Procedure: AF Ablation without contact force information — Ablation procedure will be done using TactiCath Quartz ablation catheter which can measure the amount of contact force being used. Researcher will not be made aware of contact force data when performing procedure.

SUMMARY:
The purpose of this study is to collect information about the success rate of atrial fibrillation (AF) ablation procedures using the contact force data from the TactiCath Quartz ablation catheter.

DETAILED DESCRIPTION:
Atrial fibrillation is a condition in which the upper chambers of the heart (the atria) begin to quiver (shake rapidly with small movements) instead of beating in a normal rhythm. This condition can cause blood to remain in the atria instead of moving to the lower heart chambers. AF can cause a number of other health problems and can decrease your quality of life.

Treatments for AF can include surgery, implantable devices, ablation and medication, to name a few. An ablation is a procedure that creates scar tissue in the heart to interrupt irregular heart rhythms and prevent them from coming back. The ablation procedure uses tools called catheters to treat the AF. Ablation catheters are thin, flexible plastic tubes that use electrical energy to create scars in the heart.

The amount of force applied to the heart tissue where the catheter touches (called the contact force) might help determine the success of the ablation procedure. This study would help to determine whether or not the contact force makes a difference in an effective ablation. You will be tested on both sides, at the end of the procedure to see if any problem persists.

Participants will be in this study for about 3 months. All visits in this study will correspond to standard of care visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an initial AF ablation procedure
* Able to sign informed consent and complete the 3 month follow up

Exclusion Criteria:

* Severe COPD and is unable to receive adenosine therapy during the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are undergoing an intial AF ablation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rates of dormant conduction | intraoperative
  Comparison of rates between pulmonary veins where the contact force information was known to researcher during ablation procedure versus contact force information NOT known during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States